CLINICAL TRIAL: NCT02268045
Title: A Randomized, Double-blind, Phase III Study Comparing Biosimilar Rituximab (RTXM83) Plus CHOP Chemotherapy Versus a Reference Rituximab Plus CHOP (R-CHOP) in Patients With Diffuse Large B-cell Lymphoma (DLBCL) Given as First Line
Brief Title: Study of RTXM83 Plus CHOP Chemotherapy Versus a Rituximab Plus CHOP Therapy in Patients With Non Hodgkin's Lymphoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: mAbxience Research S.L. (Industry)
Collaborators: Pisa® Farmacéutica (Unknown); Laboratorios de Productos Éticos C.E.I.S.A. (Unknown); Laboratorio Elea Phoenix S.A. (Industry); Tecnoquimicas S.A (Unknown); Innogene Kalbiotech Pte. Ltd (Industry); Libbs Farmacêutica LTDA (Industry); Key Oncologics (Pty) Ltd (Unknown); Nanolek LLC (Other); Actoverco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RTXM83-AC-01-11
Record Dates: First submitted 2014-09-19; First posted 2014-10-20 (Estimated); Results first posted 2019-09-26 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-08

CONDITIONS: Diffuse Large B-cell Lymphoma
Keywords: Non-Hodgkin Lymphoma; DLBCL; Diffuse large b-cell lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin | interventions — Rituximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RTXM83 (Experimental): Active Ingredient: Rituximab (Biosimilar)
  Interventions: Biological: RTXM83
- MabThera (Active Comparator): Active Ingredient: Rituximab
  Interventions: Biological: Mabthera

INTERVENTIONS:
Biological: RTXM83 — Rituximab biosimilar (RTXM83) will be administered in combination with CHOP chemotherapy regimen (Cyclophosphamide 750 mg/m2, Doxorubicin 50 mg/m2 and Vincristine 1.4 mg/m2 up to a maximum of 2 mg on Day 1 plus Prednisone 40 mg/m2 or 100 mg per day from Day 1 to 5) at a dose of 375 mg/m2 on Day 1 of each 3 week cycle, for 6 cycles, although the administration of 2 additional cycles may be allowed.
  Other Names: Rituximab Biosimilar
  Arms: RTXM83
Biological: Mabthera — Mabthera will be administered in combination with CHOP chemotherapy regimen (Cyclophosphamide 750 mg/m2, Doxorubicin 50 mg/m2 and Vincristine 1.4 mg/m2 up to a maximum of 2 mg on Day 1 plus Prednisone 40 mg/m2 or 100 mg per day from Day 1 to 5) at a dose of 375 mg/m2 on Day 1 of each 3 week cycle, for 6 cycles, although the administration of 2 additional cycles may be allowed.
  Other Names: Reference rituximab
  Arms: MabThera

SUMMARY:
This is a multicenter, double-blind, randomized study comparing the efficacy, pharmacokinetics (PK)/pharmacodynamics (PD), safety and immunogenicity profile of RTXM83 (rituximab biosimilar) vs reference rituximab (MabThera®), both with CHOP, as first-line treatment of Diffuse-Large-B-Cell-Lymphoma (DLBCL).

Rituximab biosimilar and MabThera® were both administered intravenously on Day 1 of each 3-week cycle with CHOP chemotherapy for six cycles. Two additional cycles of treatment were permitted at the Investigator's discretion. Patients were followed up for 9 months after last study dose.

DETAILED DESCRIPTION:
The primary endpoint of the investigation is to determine if the response rate obtained with RTXM83 combined with CHOP is non inferior to the response rate obtained with reference rituximab combined with CHOP.

The present study is a non inferiority trial and the study hypothesis is the following: H0: pc ≥ pe + δ vs. H1: pc < pe + δ where, pe: proportion of successes in the experimental group (RTXM83+CHOP) pc: proportion of successes in the control group (Reference Rituximab+CHOP) Type I error: the difference pc-pe is less than δ when in fact the difference is greater than or equal to δ ie, the investigators choose the experimental treatment when the control treatment is actually substantially better.

Type II error: the difference -pe is greater than or equal to δ when it is actually lest than δ ie, the investigators choose the control treatment when the experimental treatment is essentially just as good.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with measurable disease defined as existence of a unidimensional or bidimensional lesion greater than 2 cm in its longest diameter or malignant lymphocytosis greater than 5x109/L. Any other procedure for measurable disease in particular cases, may be allowed upon Sponsor approval
2. Newly diagnosed patients with a confirmed pathologic diagnosis of Diffuse large B cell-non-Hodgkin's lymphoma (DLBCL) with untreated CD20+ receptor (CD20+). Defined by the local Haematopathologist at the local laboratory according to World Health Organization (WHO) criteria
3. Stage II-III or IV or stage I with bulk defined by the referring physician on the basis of the Cotswolds modification of the Ann Arbor classification 2
4. Age-adjusted International Prognostic Index (IPI) score 0 or 1
5. Age ≥18 to ≤65 years of age
6. Performance status according to Eastern Cooperative Oncology Group (ECOG) of ≤2
7. Written informed consent obtained before starting any study-specific procedure
8. Females of child-bearing potential must test negative on standard serum pregnancy test and must be willing to practice appropriate contraceptive methods for the duration of the study (e.g. oral contraceptive, double barrier method, intra-uterine device, intra-muscular contraceptive)
9. All male patients must take adequate contraceptive precautions during the course of the study

Exclusion Criteria:

1. Life expectancy of less than three months
2. Any other lymphoma other than CD20+ DLBCL
3. Indolent lymphoma, Primary central nervous system (CNS) Lymphoma or gastro-intestinal Mucosa Associated Lymphoid Tissue (MALT) Lymphoma
4. Known hypersensitivity to active ingredients, excipients and murine and foreign proteins
5. Concurrent disease or general status that would exclude giving the treatment as outlined in the protocol
6. Active uncontrolled infection requiring systemic treatment with antibiotics or antiviral agents at Screening or history of documented recurrent clinically significant infection (e.g. 2 or more viral, bacterial or fungal infections requiring inpatient treatment)
7. Cardiac contra-indication to Doxorubicin therapy: non-compensated heart failure, dilated cardiomyopathy, coronary heart disease with ST segment depression on electrocardiogram (ECG), myocardial infarction in the last 6 months
8. Neurologic contra-indication to Vincristine as it is indicated in the Summary of Product Characteristics (SmPC): (e.g. peripheral neuropathy)
9. Chronic lung disease with hypoxemia measured by pulse oximetry (gasometry is not mandatory)
10. Severe uncontrolled hypertension, despite optimal medical treatment
11. Severe uncontrolled diabetes mellitus, despite optimal medical treatment
12. Renal insufficiency (Serum Creatinine >2 x Upper Normal Limit [UNL])
13. Hepatic insufficiency: aspartate aminotransferase (AST)/ alanine aminotransferase (ALT)>3 x UNL or >5 x UNL with involvement of the liver, total bilirubin >34.2 µmol/L, or both) not related to lymphoma
14. Clinical signs of cerebral dysfunction
15. Severe psychiatric disease
16. Known human immunodeficiency virus (HIV) infection or active chronic hepatitis B or C
17. Abnormal bone marrow function (platelets <100x109/L, neutrophils <1.5x109/L and Haemoglobin <9g/dL)
18. Post-transplantation lymphoproliferative disease
19. Pregnant or lactating women or women that intend to get pregnant during study or within 12 months following the last infusion
20. Treatment with any investigational product in the 30 days period before inclusion in the study
21. Prior radiotherapy to treat the DLBCL Non-Hodgkin's Lymphoma (NHL)
22. Limitation of the patient's ability to comply with the treatment or follow-up protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Actual)
Dates: Start 2013-05; Primary Completion 2016-05 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susana Millán, Phd, Study Director — mAbxience Research S.L.
Locations (87):
- Argentina (17):
  - Hosp. Interzonal "R" Carrillo, Ciudadela, Bariloche
  - Clinica Radiologica del Sur, Cipolletti, Río Negro Province
  - Clinica Viedma, Viedma, Río Negro Province
  - Hospital Britanico, Buenos Aires
  - Hospital Gral. de Agudos Donación Francisco Santojanni, Buenos Aires
  - Instituto Roffo, Buenos Aires
  - Centro Oncologico Riojano Integral (CORI), Córdoba
  - Hospital Nacional de Clinicas, Córdoba
  - Hospital Privado de Cordoba, Córdoba
  - Sanatorio Allende, Córdoba
  - Ctr. Oncologico de Rosario, Rosario
  - Inst. Cardiovascular Rosario, Rosario
  - Instituto de Hematología y Medicina Clínica Dr. Rubén Dávoli, Rosario
  - Sanatorio Parque, Rosario
  - Hospital Angel Padilla, San Miguel de Tucumán
  - Fundación ARS Médica, San Salvador de Jujuy
  - Hospital J. B. Iturraspe, Santa Fe
- Brazil (22):
  - Hospital de Caridade de Ijuí, Ijuí, Rio Grande do Sul
  - Hospital da Cidade de Passo Fundo, Passo Fundo, Rio Grande do Sul
  - Hospital São Lucas da PUCRS, Porto Alegre, Rio Grande do Sul
  - Hospital Clinicas Porto Alegre, Pôrto Alegre, Rio Grande do Sul
  - Hospital Santa Marcelina, Itaquera, São Paulo
  - Hospital Amaral Carvalho Jaú, Jaú, São Paulo
  - Hospital das Clínicas da Faculdade de Medicina de Ribeirão Preto da Universidade de São Paulo-HCFMRP, Ribeirão Preto, São Paulo
  - CEPHO - Centro de Estudos e Pesquisas de Hematologia e Oncologia / Faculdade de Medicina do ABC, Santo André, São Paulo
  - Fundação Antônio Prudente - AC Camargo Câncer Center, São Paulo, São Paulo
  - Hospital das Clinicas-UFMG, Belo Horizonte
  - UNICAMP-Univ Zeferino Vaz, Campinas
  - Hospital Uniao Oeste Paranaense de Estudos e Comabte ao Cancer (UOPECCAN), Cascavel
  - Hospital Erasto Gaertner CEPEP, Curitiba
  - Hospital das Clínicas da Universidade Federal de Goiás, Goiânia
  - Santa Casa de Porto Alegre, Porto Alegre
  - Hospital Universitário Clemente Fraga Filho - UFRJ, Rio de Janeiro
  - Instituto COI de Educação e Pesquisa, Rio de Janeiro
  - Instituto Est. de Hematologia Arthur de Siqueira Cavalcanti, Rio de Janeiro
  - Monte Tabor - Hospital São Rafael, Salvador
  - Hospital de Base de São José, São José do Vale do Rio Preto
  - Centro de Pesquisa do Instituto Brasileiro de Controle do Câncer - IBCC, São Paulo
  - Hospital Clinica Faculdade Medicina USP, São Paulo
- Colombia (3):
  - Inst. Nacional de Cancerologia, Bogotá
  - Fundación Valle de Lili, Cali
  - Hospital Pablo Tobon Uribe, Medellín
- India (12):
  - Srinivasam Cancer Care Hospital, Bangalore
  - Cancer Institute, Chennai
  - Rajiv Gandhi Cancer Institute and Research Centre, Delhi
  - Bibi General Hospital&Canc Ct, Hyderabad
  - Birla Cancer Center - SMS Hospital, Jaipur
  - Health Point Multi-specialty Hospital, Kolkata
  - Institute of Hematology and Transfusion Medicine, Kolkata
  - Netaji Subhash Chandra Bose Cancer Research Institute, Kolkata
  - Acharya Tulsi Regional Cancer Treatment and Research Institute, Madurai
  - Guru Hospital, Madurai
  - Meenakshi Mission Hospital, Madurai
  - Kailash Cancer Hospital and Research Centre, Vadodara
- Indonesia (2):
  - Dr. Hasan Sadikin Hospital, Bandung
  - Dharmais N. C. Center, Jakarta
- Imam Khomeini Complex Hospital - Cancer Institute, Tehrān, Iran
- Malaysia (4):
  - Hospital Sultanah Aminah, Johor Bahru
  - University Malaya Medical Centre - UMMC, Kuala Lumpur
  - Mount Miriam Cancer Hospital, Pulau Pinang
  - Hospital Pulau Pinang, Pulau Pinang
- Insituto Nacional de Cancerología, Mexico City, Mexico
- Instituto Privado de Hematologia e Investigaciona Clinica, Asunción, Paraguay
- Philippines (5):
  - Cebu Doctors University Hospital, Cebu
  - Perpetual Succour Hospital, Cebu
  - Davao Doctors Hospital, Davao City
  - National Kidney and Transplant Institute, Quezon City
  - Veterans Memorial Medical Center, Quezon City
- Russia (15):
  - Arkhangelsk Clinical Oncology Dispensary, Arkhangelsk
  - Kursk regional clinical oncology dispensary, Kursk
  - N.N. Blokhin Russian Cancer Research Cente, Moscow
  - National Medical Surgical Center n.a. N.I. Pirogov, Moscow
  - Murmansk regional oncology dispensary, Murmansk
  - State Budgetary Healthcare Institution of Stavropol region "Pyatigorsk oncology center", Pyatigorsk
  - Rostov Scientific Research Oncology Institute, Rostov-on-Don
  - Russian Research Center for Radiology and Surgical Technologies, Saint Petersburg
  - Saint-Petersburg State Budgetary Institution "City Clinical Oncology Dispensary", Saint Petersburg
  - Scientific Research Institute of Oncology n.a. N.N. Petrov, Saint Petersburg
  - Oncology Center # 2, Sochi
  - Komi Republican Oncology Dispensary, Syktyvkar
  - State Healthcare Institution of Tula region "Tula regional clinical hospital", Tula
  - Republican Clinical Oncology Dispensary, Ufa
  - Volgograd Regional Clinical Oncology Center, Volgograd
- South Africa (4):
  - Tygerberg Academic Hosp, Cape Town
  - Rainbow Oncology Centre, eManzimtoti
  - GVI Oncology, Port Elizabeth
  - Chris Hani Baragwanath Hospital, Soweto

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: An additional cohort of 16 patients was added (as per Iran local regulatory requirements) to the planned sample of 256 patients. The extension cohort of Iran was only considered for safety analysis.
Groups:
- RTXM83: Rituximab biosimilar (RTXM83) was administered in combination with CHOP chemotherapy regimen (Cyclophosphamide 750 mg/m2, Doxorubicin 50 mg/m2 and Vincristine 1.4 mg/m2 up to a maximum of 2 mg on Day 1 plus Prednisone 40 mg/m2 or 100 mg per day from Day 1 to 5) at a dose of 375 mg/m2 on Day 1 of each 3 week cycle, for 6 cycles. Administration of 2 additional cycles was allowed as per Investigator's criteria.
- MabThera: MabThera was administered in combination with CHOP chemotherapy regimen (Cyclophosphamide 750 mg/m2, Doxorubicin 50 mg/m2 and Vincristine 1.4 mg/m2 up to a maximum of 2 mg on Day 1 plus Prednisone 40 mg/m2 or 100 mg per day from Day 1 to 5) at a dose of 375 mg/m2 on Day 1 of each 3 week cycle, for 6 cycles. Administration of 2 additional cycles was allowed as per Investigator's criteria.
Period: Overall Study
Arm/Group | RTXM83 | MabThera
Started | 136 | 136
Completed | 120 | 116
Not Completed | 16 | 20
Not completed — Death | 4 | 4
Not completed — Disease Progression | 2 | 1
Not completed — Adverse Event | 7 | 7
Not completed — Withdrawal by Subject | 2 | 6
Not completed — Physician Decision | 0 | 1
Not completed — Protocol Violation | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- RTXM83-CHOP: Patients treated with Rituximab biosimilar in combination with CHOP chemotherapy
- MabThera-CHOP: Patients treated with Rituximab in combination with CHOP chemotherapy
- Total: Total of all reporting groups
Arm/Group | RTXM83-CHOP | MabThera-CHOP | Total
Number analyzed (Participants) | 136 | 136 | 272
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 49.0 [40.0 to 57.0] | 51.0 [41.0 to 59.0] | 51.0 [40.0 to 58.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 59 | 117
  Male | 78 | 77 | 155
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 2 | 7
  Asian | 50 | 53 | 103
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 3 | 9
  White | 75 | 78 | 153
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Initial disease stage (Ann Arbor Staging) [Count of Participants; unit: Participants] — The stage depends on both the place where the malignant tissue is located and on systemic symptoms due to the lymphoma. Ann Arbor Stage=I: Best condition; Ann Arbor Stage=IV: Worst condition
  Stage I: cancer located in a single region; Stage II: cancer located in 2 separate regions that are confined to one side of the diaphragm; Stage III: cancer spreading to both sides of the diaphragm; Stage IV: diffuse or disseminated involvement of one or more extralymphatic organs.
  Participants
    Stage I (with bulky) | 19 | 19 | 38
    Stage II | 64 | 53 | 117
    Stage III | 30 | 32 | 62
    Stage IV | 23 | 32 | 55
Presence of extra nodal lesions [Count of Participants; unit: Participants]
  No | 88 | 81 | 169
  Yes | 48 | 55 | 103
Performance Status according to Eastern Cooperative Oncology Group (ECOG) [Count of Participants; unit: Participants] — Measure Description: ECOG=0: Fully active, able to carry on all pre-disease performance without restriction; ECOG =1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature;
  Participants
    0 | 84 | 84 | 168
    1 | 52 | 50 | 102
    Missing data | 0 | 2 | 2
Age-adjusted International Prognostic Index (IPI) [Count of Participants; unit: Participants] — Age-adjusted IPI is a simplified index for comparing patients within an age group (i.e. 60 or younger, or over 60) and includes the evaluation of 3 clinical factors: Ann Arbor stage III or IV disease; ECOG performance status >=2 and ; increased serum lactate dehydrogenase levels.
  The sum of the points allotted correlates with the following risk groups:
  Low risk (0 points) - 5-year survival of 83%; Low-intermediate risk (1 point) - 5-year survival of 69%; High-intermediate risk (2 points) - 5-year survival of 46%; High risk (3 points) - 5-year survival of 32%.
  Participants
    0 | 48 | 50 | 98
    1 | 85 | 79 | 164
    2 | 3 | 7 | 10

OUTCOME MEASURES:

1. Primary Outcome: Response Rate (RR) Achieved After Cycle 6 With RTXM83 Plus CHOP Compared to the RR Obtained With Mabthera® Plus CHOP (R-CHOP) in Patients With DLBCL
Description: Per International Working Group (IWG) revised criteria for Malignant Lymphomas (Cheson et al. 2007) and assessed by positron-emission tomography scan, or by computed tomography scan and/or magnetic resonance imaging if Positron Emission Tomography (PET) scan was not feasible. Tumor response was classified according to the International Working Group criteria, as Complete Remission (CR): Complete disappearance of all detectable clinical evidence of disease and disease-related symptoms if present before therapy; Partial Response (PR): At least a 50% decrease in sum of the product of the diameters of up to six of the largest dominant nodes or nodal masses; Stable disease (SD) or; Progressive disease. Response rate was the sum of CR and PR.
Time Frame: Tumor response assessed after Cycle 6 or at the end of treatment
Population: The Intent-to-treat (ITT) population and the Per Protocol (PP) population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RTXM83-CHOP | MabThera-CHOP
Number analyzed (Participants) | 122 | 117
percentage of participants
  ITT : Response rate (CR+PR) | 83.6 [75.8 to 89.7] | 82.9 [74.8 to 89.2]
  PP : Response rate (CR+PR): number analyzed (Participants) | 111 | 104
  PP : Response rate (CR+PR) | 84.7 [76.6 to 90.8] | 81.7 [72.9 to 88.6]
Statistical Analysis 1: Comparison: RTXM83-CHOP vs MabThera-CHOP; Test type: Non-Inferiority or Equivalence — The RR, with the corresponding 95% CI, was calculated for each treatment arm and compared using Fisher's exact test at a one-sided 0.025 type I error rate. A non-inferiority margin of 13% was assumed with ≥ 80% power to detect treatment differences. Non-inferiority was concluded if the one-sided 95% CI was above the -13% margin set for the study; Percentage difference = 0.7, 95% CI 1-sided [lower limit -13] — For the ITT population
Statistical Analysis 2: Comparison: RTXM83-CHOP vs MabThera-CHOP; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; percentage difference = 3, 95% CI 1-sided [lower limit -13] — For the PP population

2. Secondary Outcome: AUC 0-∞ (h μg/mL) at Cycle 1 of RTXM83 and Mabthera®
Description: Compare the pharmacokinetic (PK) parameter (AUC 0-∞) calculated from start of the first infusion until start of the second infusion (i.e. at Cycle 1) in a population PK model.
  For the PK similarity assessments, regulatory guidelines on bioequivalence were followed whereby two treatments are judged not to be different from one another if the 90% confidence interval (CI) of the ratio between the geometric means of the measure (AUC 0-∞ ) falls completely within the range 80%-125%.
Time Frame: Cycle 1 (first dose): Day 1 (pre-dose, mid-infusion), Day 8 and Day 15
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: ng.h/mL
Groups:
- RTXM83-CHOP: Patients treated with Rituximab biosimilar with CHOP chemotherapy
- MabThera- CHOP: Patients treated with Rituximab in combination with CHOP chemotherapy
Arm/Group | RTXM83-CHOP | MabThera- CHOP
Number analyzed (Participants) | 127 | 123
ng.h/mL | 44519 (32) | 44874 (47)
Statistical Analysis 1: Comparison: RTXM83-CHOP vs MabThera- CHOP; Test type: Equivalence — Two treatments are judged not to be different from one another if the 90% CI of the ratio of a log-transformed exposure measure (AUC) falls completely within the range 80%-125%; ratio RTXM83 to Mabthera = 99.2, 90% CI 2-sided [93.6 to 105] — For the ratio: RTXM83 represents the numerator and Mabthera the denominator

3. Secondary Outcome: AUC 0-∞ (h μg/mL) at Cycle 6 of RTXM83 and Mabthera®
Description: Compare the PK parameter (AUC 0-∞) calculated from start of the first infusion until Day 21 of administration of Cycle 6 in a population PK model.
  For the PK similarity assessments, regulatory guidelines on bioequivalence were followed whereby two treatments are judged not to be different from one another if the 90% confidence interval (CI) of the ratio between the geometric means of the measure (AUC 0-∞ ) falls completely within the range 80%-125%.
Time Frame: Cycle 6 (last dose): Day 1, Day 8, Day 15 and Day 21
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: ng.h/mL
Arm/Group | RTXM83-CHOP | MabThera- CHOP
Number analyzed (Participants) | 113 | 105
ng.h/mL | 60875 (22) | 59079 (40)
Statistical Analysis 1: Comparison: RTXM83-CHOP vs MabThera- CHOP; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; ratio RTXM83 to Mabthera = 103, 90% CI 2-sided [98.5 to 107] — For the ratio: RTXM83 represents the numerator and Mabthera the denominator

4. Secondary Outcome: Cmax (μg/mL) at Cycle 1 of RTXM83 and Mabthera®
Description: Compare the PK parameter (Cmax) calculated from start of the first infusion until start of the second infusion (i.e. at Cycle 1) in a population PK model.
  For the PK similarity assessments, regulatory guidelines on bioequivalence were followed whereby two treatments are judged not to be different from one another if the 90% confidence interval (CI) of the ratio between the geometric means of the measure (Cmax) falls completely within the range 80%-125%.
Time Frame: Cycle 1 (first dose): Day 1 (pre-dose, mid-infusion), Day 8 and Day 15
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | RTXM83-CHOP | MabThera- CHOP
Number analyzed (Participants) | 127 | 123
μg/mL | 196.8 (24) | 197.5 (31)
Statistical Analysis 1: Comparison: RTXM83-CHOP vs MabThera- CHOP; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; ratio RTXM83 to Mabthera = 99.6, 90% CI 2-sided [93.9 to 105] — For the ratio: RTXM83 represents the numerator and Mabthera the denominator

5. Secondary Outcome: Cmax (μg/mL) at Cycle 6 of RTXM83 and Mabthera®
Description: Compare the PK parameter (Cmax) calculated from start of the first infusion until Day 21 of administration of Cycle 6 in a population PK model.
  For the PK similarity assessments, regulatory guidelines on bioequivalence were followed whereby two treatments are judged not to be different from one another if the 90% confidence interval (CI) of the ratio between the geometric means of the measure (AUC 0-∞ ) falls completely within the range 80%-125%.
Time Frame: Cycle 6 (last dose): Day 1, Day 8, Day 15 and Day 21
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | RTXM83-CHOP | MabThera- CHOP
Number analyzed (Participants) | 113 | 105
μg/mL | 291 (21) | 279 (36)
Statistical Analysis 1: Comparison: RTXM83-CHOP vs MabThera- CHOP; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; ratio RTXM83 to Mabthera = 104, 90% CI 2-sided [99.5 to 109] — For the ratio: RTXM83 represents the numerator and Mabthera the denominator

6. Secondary Outcome: Percentage Change From Baseline in Pharmacodynamic (PD) Markers (CD19+ and CD20+ Cells) Blood Counts of RTXM83 and Mabthera®
Description: CD19 and CD20 are proteins found on the cell surface of B cells, and they can be detected in peripheral blood by flow cytometry. Flow cytometry of peripheral blood was performed for immediate analysis of cells with cluster of differentiation 19 (CD19+) and CD20+.
  To compare the percent Change From Baseline ((Cycle 1 pre-dose) in pharmacodynamic markers (CD19+ and CD20+ Cells) in Peripheral Blood achieved in RTXM83 and Mabthera® arms at Cycle 1 end of infusion (EOI), 6 months and 9 months after last dose of treatment.
Time Frame: Up to follow-up 3 (FU3); 9 months after last dose of treatment
Population: Data were provided for the number of samples available at each visit.
Measure: Median (Full Range); unit: percentage change in cells
Arm/Group | RTXM83-CHOP | MabThera- CHOP
Number analyzed (Participants) | 77 | 74
percentage change in cells
  Cycle 1 EOI, CD19+ | -96.8 [-100 to 10] | -94.6 [-100 to 525]
  At 6 months after last dose, CD19+: number analyzed (Participants) | 61 | 50
  At 6 months after last dose, CD19+ | -95.7 [-100 to 833] | -98.3 [-100 to 4380]
  At 9 months after last dose, CD19+: number analyzed (Participants) | 60 | 50
  At 9 months after last dose, CD19+ | -33 [-100 to 13600] | -42.3 [-100 to 10300]
  Cycle 1 EOI, CD20+: number analyzed (Participants) | 76 | 71
  Cycle 1 EOI, CD20+ | -100 [-100 to -16.7] | -100 [-100 to 7400]
  At 6 months after last dose, CD20+: number analyzed (Participants) | 60 | 51
  At 6 months after last dose, CD20+ | -98.9 [-100 to 700] | -100 [-100 to 6990]
  At 9 months after last dose, CD20+: number analyzed (Participants) | 59 | 51
  At 9 months after last dose, CD20+ | -22.2 [-100 to 69100] | -30.6 [-100 to 12400]

7. Secondary Outcome: Comparable Safety Profile in Both Treatment Arms
Description: Compare the frequency and severity of treatment emergent adverse events (TEAEs) and serious adverse events (SAEs) reported in each treatment arm.
Time Frame: Up to FU3; 9 months after last dose of treatment
Population: All patients receiving at least one dose of the study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | RTXM83-CHOP | MabThera-CHOP
Number analyzed (Participants) | 136 | 136
Participants
  At least one TEAE (any causality) | 131 | 131
  At least one grade 3/4 TEAE (any causality) | 75 | 80
  TEAEs related to treatment | 125 | 119
  Serious TEAEs (any causality) | 47 | 45
  TEAE led to drug discontinuation (any causality) | 6 | 7

8. Secondary Outcome: Comparable Immunogenicity Profile Between RTXM83 and Mabthera®
Description: Anti-Drug Antibody (ADA) developed de novo (seroconversion) after 6 cycles of treatment and 9 months of follow-up.
Time Frame: Up to FU3; 9 months after last dose of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | RTXM83-CHOP | MabThera-CHOP
Number analyzed (Participants) | 127 | 125
Participants
  Seroconversion | 3 | 4
  No seroconversion | 124 | 121

9. Secondary Outcome: Event Free Survival (EFS) in RTXM83 Arm and Mabthera® Arm
Description: Time from randomization to any of the following events: progressive disease, no achievement of CR, PR associated with treatment in excess of that per protocol, SD, relapse after achievement of CR, or death from any cause, whichever comes first.
Time Frame: Up to FU3; 9 months after last dose of treatment
Population: Number of patients with an EFS event (progressive disease, no achievement of CR, PR associated with treatment more than that per protocol, stable disease, relapse after achievement of CR, or death from any cause, whichever comes first).
Measure: Median (95% Confidence Interval); unit: time (months)
Arm/Group | RTXM83-CHOP | MabThera- CHOP
Number analyzed (Participants) | 122 | 117
time (months) | 12.5 [4.4 to NA] — Upper limit of the Confidence Interval was not achieved due to short time follow up | 8.6 [4.6 to NA] — Upper limit of the Confidence Interval was not achieved due to short time follow up
Statistical Analysis 1: Comparison: RTXM83-CHOP vs MabThera- CHOP; Test type: Other; p = 0.4570, Log Rank

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the study start, during the study and up to 30 days after the end of study treatment.
Description: Graded according to the National Cancer Institute-Common Toxicity Criteria (NCI-CTC; version 4.0) and categorized using the MedDRA (version 16.0) terminology.
Arm/Group | RTXM83-CHOP | MabThera-CHOP
All-Cause Mortality (participants affected / at risk) | 8/136 | 12/136
Serious Adverse Events (participants affected / at risk) | 47/136 | 45/136
Other Adverse Events (participants affected / at risk) | 131/136 | 131/136
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RTXM83-CHOP (N=136) | MabThera-CHOP (N=136)
Neutropenia (Blood and lymphatic system disorders) | 10 | 8
Leukopenia (Blood and lymphatic system disorders) | 6 | 5
Diarrhoea (Gastrointestinal disorders) | 4 | 3
Pyrexia (General disorders) | 5 | 5
Pneumonia (Infections and infestations) | 6 | 5
Septic shock (Infections and infestations) | 3 | 3
Lung infection (Infections and infestations) | 2 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 19 | 7
Dehydration (Metabolism and nutrition disorders) | 3 | 3
Hyponatremia (Metabolism and nutrition disorders) | 3 | 3
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 2 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | RTXM83-CHOP (N=136) | MabThera-CHOP (N=136)
Neutropenia (Blood and lymphatic system disorders) | 53 | 59
Anaemia (Blood and lymphatic system disorders) | 44 | 39
Leukopenia (Blood and lymphatic system disorders) | 37 | 38
Febrile Neutropenia (Blood and lymphatic system disorders) | 21 | 11
Lymphopenia (Blood and lymphatic system disorders) | 10 | 14
Thrombocytopenia (Blood and lymphatic system disorders) | 9 | 11
Nausea (Gastrointestinal disorders) | 35 | 42
Vomiting (Gastrointestinal disorders) | 23 | 27
Diarrhoea (Gastrointestinal disorders) | 24 | 24
Constipation (Gastrointestinal disorders) | 17 | 18
Abdominal Pain (Gastrointestinal disorders) | 16 | 13
Stomatitis (Gastrointestinal disorders) | 12 | 14
Abdominal pain upper (Gastrointestinal disorders) | 9 | 11
Pyrexia (General disorders) | 29 | 23
Fatigue (General disorders) | 14 | 22
Asthenia (General disorders) | 19 | 16
Oedema peripheral (General disorders) | 8 | 5
Chills (General disorders) | 3 | 7
Pneumonia (Infections and infestations) | 8 | 8
Urinary tract infection (Infections and infestations) | 5 | 7
Oral candidiasis (Infections and infestations) | 1 | 7
Blood lactate dehydrogenase increased (Investigations) | 8 | 11
Weight decreased (Investigations) | 9 | 9
Gamma-glutamyltransferase increased (Investigations) | 2 | 10
Hypokalaemia (Metabolism and nutrition disorders) | 12 | 13
Hypocalcaemia (Metabolism and nutrition disorders) | 12 | 8
Decreased appetite (Metabolism and nutrition disorders) | 10 | 9
Hyperglycaemia (Metabolism and nutrition disorders) | 8 | 10
Hyponatraemia (Metabolism and nutrition disorders) | 8 | 8
Dyslipidaemia (Metabolism and nutrition disorders) | 7 | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 7 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 9
Myalgia (Musculoskeletal and connective tissue disorders) | 7 | 5
Neuropathy peripheral (Nervous system disorders) | 26 | 13
Headache (Nervous system disorders) | 14 | 17
Paraesthesia (Nervous system disorders) | 14 | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 16 | 13
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 | 6
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 | 5
Alopecia (Skin and subcutaneous tissue disorders) | 35 | 27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No